CLINICAL TRIAL: NCT02101866
Title: A Randomized, Single-Center, Open-Label, Two-Period, Two-Sequence, Crossover, Comparative Study to Compare the Oral Bioavailability of Single Doses of Two Vapendavir Drug Product Formulations in Healthy Volunteers
Brief Title: A Study to Compare the Oral Bioavailability of Single Doses of Two Vapendavir Drug Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biota Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Vaxart (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BTA798-103
Record Dates: First submitted 2014-03-24; First posted 2014-04-02 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Healthy
Keywords: Bioavailability Study; Aviragen Therapeutics, Inc.; Aviragen Therapeutics; Aviragen
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vapendavir 300 mg tablet (Experimental): Vapendavir 300 mg tablet single dose with up to 7 day washout period followed by two vapendavir 132 mg capsules single dose
  Interventions: Drug: Vapendavir 300 mg tablet
- Two Vapendavir 132 mg capsules (Experimental): Two Vapendavir 132 mg capsules single dose with up to 7 day washout period followed by Vapendavir 300 mg tablet single dose
  Interventions: Drug: Vapendavir 132 mg capsules

INTERVENTIONS:
Drug: Vapendavir 300 mg tablet — tablet - single dose
  Arms: Vapendavir 300 mg tablet
Drug: Vapendavir 132 mg capsules — 2 capsules - single dose
  Arms: Two Vapendavir 132 mg capsules

SUMMARY:
This Phase 1 study aims to determine the oral bioavailability of a single dose of a new vapendavir tablet formulation and compare it to that of the previous vapendavir capsule formulation. The safety of both drug products will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Must be male or female between 18 and 55 years of age (inclusive) with BMI between 18 and 30 kg/m2 (inclusive), and weight ≥50 kg at the time of screening
* Capable of giving written informed consent
* Subject is able to understand and comply with the protocol requirements, instructions and restrictions
* Healthy on the basis of physical examination, medical history, medication usage, VS, ECGs, and clinical laboratory tests
* Female subjects must be of non-childbearing potential
* Male subjects must agree to use a double barrier method of birth control

Exclusion Criteria:

* Positive results for Hepatitis B, Hepatitis C, or HIV
* Frequent use of tobacco products, including cigarettes, cigars, chewing tobacco
* A medical history of significant hematological, gastrointestinal, respiratory, renal, hepatic, cerebrovascular, immunologic, psychiatric or cardiovascular disease or event; Current or recent respiratory infection
* Presence or history of significant allergy
* Clinically significant abnormalities noted on ECG
* Screening vital signs representing sustained elevated blood pressure
* Presence of significant gastrointestinal abnormalities
* Safety laboratory abnormalities noted at screening which are clinically significant
* Current or defined history of abuse of alcohol or illicit drugs
* A positive pregnancy test at screening
* Poor vein access or fear of venipuncture or sight of blood

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Systemic exposure profile of a single dose of a vapendavir 300 mg tablet compared to the exposure profile following a single dose of two 132 mg vapendavir capsules | maximum up to 46 days
  PK and statatistical analyses will be performed to determine the Primary Outcome Measure

CONTACTS AND LOCATIONS:
Overall Officials: Mark Matson, M.D., Principal Investigator — Prism Research, Inc
Locations (1):
- Investigative Site, Saint Paul, Minnesota, United States